CLINICAL TRIAL: NCT06284499
Title: Effect of Different Fixed Lingual Retainers on Tooth Stability
Status: Withdrawn | Type: Observational
Why Stopped: Completed
Sponsor: Mustafa Kemal University (Other)
Responsible Party: Principal Investigator, Osman Fatih Arpag, associate professor, Mustafa Kemal University
Other Study IDs: 26308819120
Record Dates: First submitted 2024-02-08; First posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Effect of Lingual Retainers on Tooth Stability
Keywords: Mobility; Lingual Retainer; Retention; Periotest®

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group 1: Group 1 (n = 31), which contained patients fitted with 0.038 × 0.016" stainless steel wire (Ortho FlexTech® chain, Reliance Orthodontic Products, Itasca, IL, USA)
  Interventions: Other: measuring tooth stability after orthodontic treatment using a Periotest® device.
- Group 2: Group 2 (n = 23), which contained patients fitted with 0.010 × 0.026" 8-braided dead soft wire (Bond-A-Braid,Reliance Orthodontic Products, Itasca, IL, USA)
  Interventions: Other: measuring tooth stability after orthodontic treatment using a Periotest® device.
- Group 3: Group 3 (n = 28), which contained patients fitted with 0.0215" 5-stranded stainless steel wire (Penta-One®, Masel Orthodontics, Carlsbad, CA, USA)
  Interventions: Other: measuring tooth stability after orthodontic treatment using a Periotest® device.
- Control group: Control group (n = 20), which contained individuals who had not received any orthodontic treatment
  Interventions: Other: measuring tooth stability after orthodontic treatment using a Periotest® device.

INTERVENTIONS:
Other: measuring tooth stability after orthodontic treatment using a Periotest® device. — The tooth mobility was determined by taking three repeat measurements from each tooth and calculating the average of these measurements, using a Periotest® device.

SUMMARY:
Objective: The aim of this study was to compare the effect of different fixed lingual retainers (LRs) on tooth stability after orthodontic treatment using a Periotest® device.

Materials and methods: A total of 82 patients (43 females and 39 males; mean age = 18.61 ± 3.71 years) with no missing teeth in the lower inter-canine region were treated with fixed orthodontic mechanics. At the completion of the orthodontic treatment, each patient was fitted with either Ortho FlexTech (Reliance; Group I), dead soft 8-braided (Bond-A-Braid, Reliance; Group II), or 5-stranded (PentaOne, Masel; Group III) LR wire. A control group consisting of people with a healthy periodontal condition and no bone loss was included (Control; Group C). The mobility of the lower anterior teeth on the right and left sides was measured using a Periotest® device before (T0), immediately after (T1), and 10 months after (T2) the application of the LR. Statistical analyses were performed using one-way ANOVA followed by post hoc LSD, repeated ANOVA with Bonferroni post hoc test, and Pearson χ2 tests.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of orthodontic treatment with optimum oral hygiene
* A duration of orthodontic treatment with fixed appliances of more than 12 months
* No missing teeth, restorations, or morphological crown anomalies
* No radiological alveolar bone loss in the mandibular inter-canine region.

Exclusion Criteria:

* Individuals with periodontal problems, such as gingival bleeding and recession, parafunctional habits (e.g., clenching and grinding),
* Any radiological pathology around the lower anterior teeth

Ages: 14 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Patients seeking orthodontic treatment in an university hospital
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-01-15 (Actual); Study Completion 2023-10-13 (Actual)

PRIMARY OUTCOMES:
Assessment of tooth stability after orthodontic lingual retainer wire application using periotest device | Up to 10 months
  Tooth mobility measured just before and after lingual retainer wire application

CONTACTS AND LOCATIONS:
Locations (1):
- Hatay Mustafa Kemal University, Faculty of Dentistry, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Littlewood SJ, Kandasamy S, Huang G. Retention and relapse in clinical practice. Aust Dent J. 2017 Mar;62 Suppl 1:51-57. doi: 10.1111/adj.12475. PMID 28297088
- [Background] Bishara SE, Treder JE, Damon P, Olsen M. Changes in the dental arches and dentition between 25 and 45 years of age. Angle Orthod. 1996;66(6):417-22. doi: 10.1043/0003-3219(1996)0662.3.CO;2. PMID 8974177
- [Background] Johnston CD, Littlewood SJ. Retention in orthodontics. Br Dent J. 2015 Feb 16;218(3):119-22. doi: 10.1038/sj.bdj.2015.47. PMID 25686428
- [Background] Golshah A, Feyli SA. Bond Strength and Deflection of Four Types of Bonded Lingual Retainers. Int J Dent. 2022 Feb 24;2022:1707520. doi: 10.1155/2022/1707520. eCollection 2022. PMID 35251180
- [Background] Kucera J, Marek I, Littlewood SJ. The effect of different bonded retainer wires on tooth mobility immediately after orthodontic treatment. Eur J Orthod. 2022 Mar 30;44(2):178-186. doi: 10.1093/ejo/cjab038. PMID 34374751
- [Derived] Kucuk EB, Celik Guler O, Fatih Arpag O, Eren HK. Effect of different fixed lingual retainers on tooth mobility: prospective clinical study. Acta Odontol Scand. 2025 Dec 10;84:577-582. doi: 10.2340/aos.v84.44808. PMID 41369988